CLINICAL TRIAL: NCT01107262
Title: Avian Influenza Studies In Lebanon
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: AVIFLU -XPD09-010
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2011-10-27 (Estimated); Status verified 2011-10

CONDITIONS: Avian Influenza; Virus Diseases
Keywords: H5N1 Subtype; Avian viruses; Highly pathogenic avian influenza (HPAI)
MeSH Terms: conditions — Influenza in Birds; Virus Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — A trained phlebotomist will collect a tube of blood (7.5ml) in serum separator tubes. The blood will be allowed to clot at room temperature then centrifuged on the same day. Serum specimens will be aliqouted into multiple cryovials, labelled and preserved at -20°C until ready for laboratory study.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Poultry exposed adults: This seroepidemiological study proposes to compare adults with occupational exposure to poultry with non-poultry exposed adult controls for evidence of previous infections with AI viruses.In this study, any person with occupational exposure to poultry i.e. works in poultry production facility or raises a smaller number of poultry on his/her farm will be considered exposed. The questionnaire used in this study will capture poultry exposure data through a group of variables assessing type of occupational setting, length of time of exposure, flock size, type of work performed, and personal protective equipment (PPE) used.
- Poultry Non-exposed Adult Controls: Controls, adults who were never exposed to poultry, will be enrolled from urban areas such as the capital Beirut. Controls will be invited to volunteer by word of mouth at public/community sites.

SUMMARY:
The highly pathogenic avian influenza (HPAI) H5N1 virus arrived in the Middle East in 2005 and has since established itself in local domestic birds and is now considered endemic in several Middle Eastern countries.Few studies indicate the presence of low pathogenicity avian influenza (LPAI) viruses of the H9 type among Lebanese poultry and wild birds. These studies also provide some evidence suggesting that humans exposed to these sick birds are showing elevated antibody titers against these LPAI H9 viruses.

This study will focus on the following objectives:

* To determine the seroprevalence of AI in poultry-exposed and non-exposed human populations.
* To identify risk factors associated with AI infections in occupationally-exposed poultry workers.
* To conduct nation-wide cross-sectional surveillance for AI viruses among domestic birds in low biosecurity farms and backyard flocks.

DETAILED DESCRIPTION:
This study will examine the sera of 200 poultry-exposed adults and 50 adult controls and administer questionnaires to identify risk factors for AI infections in human beings.Study volunteers will be interviewed regarding their exposures, medical history, and behaviors using a close-ended questionnaire specifically tailored for this study. A blood sample will be collected from every participant to verify presence of antibodies against the viruses under study. All study materials are in English and Arabic. Along side the human aspect of the study, specimens will be collected from the birds that the individual handles.

This study hypothesizes that they will find evidence of previous infection with these viruses among poultry workers. Furthermore, the study team will collect animal specimens from the farms of the study volunteers and determine the types of Avian Influenza viruses that they harbour.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old.
* Be willing to participate by signing a consent form, completing the study questionnaire, and providing a blood sample.

Exclusion Criteria:

* Less than 18 years old.
* Any known immunosuppressive condition or immune deficiency disease (including HIV infection), or ongoing receipt of any immunosuppressive therapy. (Note that we have chosen to exclude such populations because of their increased risk of acquiring infections, they are relatively few, and are not representative of a national sample).
* Any individual with unknown poultry exposure status, or who was exposed to poultry more than 5 years ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will be conducted in the rural areas of Lebanon where poultry production is located.Specifically, three main regions will be included in this study, the Beqaa, North Lebanon, and South Lebanon regions.The Mount Lebanon and Beirut regions are heavily urbanized and poultry production in these regions is minimal.Poultry-exposed individuals will be enrolled according to the following scheme:100 from Beqaa, 50 from North Lebanon, and 50 from South Lebanon. The 50 non-exposed individuals will be enrolled from Beirut.
  Villages will be randomly selected from each of the 3 regions where enrollment will occur.Each village will be assigned a number and then a random digit sheet will be generated and used to randomly select villages.
  Controls, adults who were never exposed to poultry, will be enrolled from urban areas such as the capital Beirut. Controls will be invited to volunteer by word of mouth at public/community sites.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The seroprevalence of Avian Influenza in poultry-exposed and non-exposed human populations. | 1 year
Risk factors associated with AI infections in occupationally-exposed poultry workers. | 1 year
Nation-wide cross-sectional surveillance for AI viruses among domestic birds in low biosecurity farms and backyard flocks. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Ghazi Kayali, Ph.D, MPH, Principal Investigator — St. Jude Children's Research Hospital
Locations (2):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States
- American University of Beirut, Beirut, Beyrouth, Lebanon

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org